CLINICAL TRIAL: NCT03472560
Title: A PHASE 2, OPEN LABEL STUDY TO EVALUATE SAFETY AND CLINICAL ACTIVITY OF AVELUMAB (BAVENCIO (REGISTERED)) IN COMBINATION WITH AXITINIB (INLYTA (REGISTERED)) IN PATIENTS WITH ADVANCED OR METASTATIC PREVIOUSLY TREATED NON-SMALL CELL LUNG CANCER OR TREATMENT NAÏVE CISPLATIN-INELIGIBLE UROTHELIAL CANCER JAVELIN MEDLEY VEGF
Brief Title: A Study of Avelumab in Combination With Axitinib In Non-Small Cell Lung Cancer (NSCLC) or Urothelial Cancer (Javelin Medley VEGF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated since there was no need for further safety or efficacy data to be collected. The participants having benefit from the Investigational treatments have been moved to a continuation study (NCT05059522)
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B9991027; 2017-004345-24 (EudraCT Number); AVE/ AXI COMBO UC (Other: Alias Study Number); AVE/AXI COMBO UC/NSCLC (Other: Alias Study Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-21 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Non-Small Cell Lung Cancer; Urothelial Cancer
Keywords: Cancer; non-small cell lung cancer; non small cell lung cancer; NSCLC; lung cancer; urothelial cancer; bladder cancer; Avelumab; Bavencio; Axitinib; Inlyta
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms | interventions — avelumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab in combination with axitinib (Experimental): Avelumab administered at 800 mg IV every two weeks in combination with axitinib, 5 mg PO BID.
  Interventions: Drug: Avelumab (MSB0010718C); Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Avelumab (MSB0010718C) — IV treatment: Avelumab administered at 800 mg IV every two weeks
  Other Names: Bavencio
Drug: Axitinib (AG-013736) — Oral treatment: Axitinib given 5 mg PO BID
  Other Names: Inlyta

SUMMARY:
This is a Phase 2 study to evaluate the safety and efficacy of avelumab in combination with axitinib in patients with advanced or metastatic non-small cell lung cancer (NSCLC) who have received at least one prior platinum containing therapy, and in treatment naïve patients with advanced or metastatic urothelial cancer, who are ineligible for cisplatin containing chemotherapy for their advanced disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (NSCLC) Cohort: Histologically or cytologically confirmed diagnosis of NSCLC that is locally advanced or metastatic; No activating EGFR mutations, ALK or ROS1 translocations/rearrangements where testing is standard of care; received at least 1 prior platinum-based chemotherapy regimen for locally advanced or metastatic NSCLC; No more than 2 prior lines of systemic therapy for locally advanced or metastatic disease (If disease progression occurred during or within 6 months after neoadjuvant/adjuvant chemotherapy or radiotherapy-chemotherapy, the regimen is counted as 1 prior treatment regimen towards the allowed limit of prior treatment regimens); Checkpoint inhibitor naïve.
* Urothelial Cancer (UC) Cohort: Histologically or cytologically confirmed diagnosis of transitional cell carcinoma (TCC) of the urothelium (if mixed, more than 50% TCC component) including bladder, urethra, ureters, or renal pelvis that is locally advanced or metastatic; No prior systemic treatment for locally advanced or metastatic disease; Prior neoadjuvant or adjuvant therapy is permitted if disease progression occurred >12 months after the completion of therapy; Checkpoint inhibitor naïve; Ineligible for receiving cisplatin-containing front-line chemotherapy based at least one of the following criteria: ECOG performance status (PS) 2; Renal dysfunction (defined as creatinine-clearance <60 ml/min); Grade 2 peripheral neuropathy; Grade 2 hearing loss (hearing loss measured by audiometry of 25 decibels at two contiguous frequencies).
* At least 1 measurable lesion by RECIST v1.1 not previously irradiated.
* Availability of an archival FFPE tumor tissue block from primary diagnosis specimen or metastatic specimen or 15 unstained slides (10 minimum). If an archived sample is not available, a fresh tumor biopsy must be performed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. For UC patients, ECOG performance 2 is permitted (cisplatin ineligibility criterion)

Exclusion Criteria:

* Prior immunotherapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-GITR, anti-LAG-3, anti-TIM-3 or anti-CTLA-4 antibody (including ipilimumab).
* Newly diagnosed brain metastases or known symptomatic brain metastases requiring steroids.
* Radiologically documented evidence of major blood vessel invasion or encasement by cancer or intratumor cavitation, regardless of tumor histology.
* Active autoimmune disease (that might deteriorate when receiving an immunostimulatory agent).
* Current use of immunosuppressive medication (except for those listed in protocol).
* Known prior severe hypersensitivity to the investigational products /monoclonal antibodies.
* Known history of immune-mediated colitis, inflammatory bowel disease, immune-mediated pneumonitis, pulmonary fibrosis.
* NCI CTCAE Grade 3 hemorrhage within 28 days prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (13):
  - Arizona Oncology Associates- Saguaro Cancer Center, Glendale, Arizona
  - Arizona Oncology Associates, Goodyear, Arizona
  - Arizona Oncology Associates- Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology Associates- Deer Valley Cancer Center, Phoenix, Arizona
  - Arizona Oncology Associates- East Valley Cancer Center, Tempe, Arizona
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Oncology Hematology Associates, Springfield, Missouri
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Hospital Cancer Center, Greenville, South Carolina
- Hungary (3):
  - Bacs-Kiskun Megyei Korhaz Onkoradiologiai Kozpont, Kecskemét
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (4):
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - Cardiologia - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - Farmacia Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - UOC di Radiologia - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
- Poland (4):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Regionalny Szpital Specjalistyczny Im. Dr. Wladyslawa Bieganskiego w Grudziadzu, Grudziądz
  - Centrum Medyczne Dom Lekarski S.A., Szczecin
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie w Warszawie, Warsaw
- Russia (4):
  - GBUZ of Stavropol Territory "Pyatigorsk Inter-regional Oncology Dispanser", Pyatigorsk, Stavropol Territory
  - LLC "University clinic of headache", Moscow
  - Limited Liability Company "VitaMed" (LLC "VitaMed"), Moscow
  - LLC "University Clinic of Headache", Moscow
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Asan Medical Center, Songpa-gu, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (2):
  - Instituto Catalan de Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon, Castellon
- Taiwan (2):
  - Chi Mei Hospital, Liouying, Tainan, Liouying District
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Galffy G, Lugowska I, Poddubskaya EV, Cho BC, Ahn MJ, Han JY, Su WC, Hauke RJ, Dyar SH, Lee DH, Serwatowski P, Estelles DL, Holden VR, Kim YJ, Vladimirov V, Horvath Z, Ghose A, Goldman A, di Pietro A, Wang J, Murphy DA, Alhadab A, Laskov M. A phase II open-label trial of avelumab plus axitinib in previously treated non-small-cell lung cancer or treatment-naive, cisplatin-ineligible urothelial cancer. ESMO Open. 2023 Jun;8(3):101173. doi: 10.1016/j.esmoop.2023.101173. Epub 2023 May 2. PMID 37141847
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991027

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with advanced or metastatic non- small cell lung cancer (NSCLC) and received at least 1 prior platinum-containing therapy or participants with advanced or metastatic urothelial cancer (UC) and were treatment naïve and ineligible for cisplatin-containing chemotherapy for their advanced disease were enrolled.
Pre-assignment Details: A total of 104 participants were screened, out of which 43 participants failed screening and 61 participants were enrolled into the study.
Groups:
- NSCLC Avelumab + Axitinib: Participants received avelumab 800 milligrams (mg) intravenous dose every two weeks, (Day 1 and 15) of each 28-day cycle in combination with axitinib 5 mg twice daily dose on a continuous dosing schedule.
- UC Avelumab + Axitinib: Participants received avelumab 800 mg intravenous dose every two weeks, (Day 1 and 15) of each 28-day cycle in combination with axitinib 5 mg twice daily dose on a continuous dosing schedule.
Period: Overall Study
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Started | 41 | 20
Completed | 0 | 0
Not Completed | 41 | 20
Not completed — Subject transfer to continuation protocol | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Progressive disease | 24 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Death | 7 | 4
Not completed — Adverse Event | 5 | 3
Not completed — Global deterioration of health status | 0 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who received at least one dose of avelumab and axitinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib | Total
Number analyzed (Participants) | 41 | 20 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (8.93) | 70.7 (8.66) | 66.16 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 30 | 12 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 40 | 17 | 57
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 1 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 17 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response- Objective Response Rate (ORR)
Description: ORR: percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR) based on investigator's assessment as per Response Evaluation Criteria in Solid Tumours (RECIST version [v] 1.1). Both CR and PR were confirmed by repeat assessments performed no less than 4 weeks after criteria for response was first met. Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<]10 millimeter [mm]). No new lesions. PR was defined as greater than or equal to (>=) 30 percent (%) decrease under baseline of sum of diameters of all target lesions. Short axis was used in sum for target nodes, while longest diameter was used in sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease was defined as not qualifying for CR, PR, Progressive Disease.
Time Frame: Baseline up to 56 months
Population: Full Analysis Set included all participants who received at least one dose of avelumab and axitinib. Participants were classified according to the study treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 20
Percentage of participants | 31.7 [18.1 to 48.1] | 10.0 [1.2 to 31.7]

2. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) During the On-Treatment Period
Description: An Adverse Event (AE) was any untoward medical occurrence attributed to study drug in a participant who received avelumab or axitinib. Treatment-emergent adverse events (TEAEs) were those events with onset dates occurring during the on-treatment period (the time from the first dose of study treatment through minimum 30 days post last dose of study treatment or start day of new anti-cancer treatment -1 day).
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment or start of new anti-cancer treatment -1 day (maximum up to 56 months)
Population: Safety analysis set included all participants who received at least one dose of study drug (avelumab or axitinib). Participants were classified according to the study treatment received.
Measure: Number; unit: Percentage of Participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 20
Percentage of Participants | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With Hematology Test Results of Maximum National Cancer Institute; Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade During the On-Treatment Period
Description: The following hematology parameters were assessed: anemia, hemoglobin increased, international normalized ratio (INR) increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased and white blood cell decreased. Laboratory abnormality events were graded according to NCI CTCAE v 4.03 (grade 3= severe and grade 4= life-threatening). Categories with non-zero values are presented.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study drug (avelumab or axitinib). Participants were classified according to the study treatment received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 18
Percentage of participants
  Lymphocyte count decreased (Grade >=3) | 12.2 | 5.6
  Neutrophil count decreased (Grade >=3) | 2.4 | 0
  Platelet count decreased (Grade >=3) | 0 | 5.6
  White blood cell decreased (Grade >=3) | 2.4 | 0

4. Secondary Outcome: Percentage of Participants With Chemistry Test Results of Maximum CTCAE Grade During the On-Treatment Period
Description: The following chemistry parameters were assessed: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, cholesterol high, creatine phosphokinase (CPK) increased, creatinine increased, gamma-glutamyl transferase (GGT) increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypertriglyceridemia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase increased and serum amylase increased. Laboratory abnormalities were graded according CTCAE version 4.03 (grade 3= severe, grade 4= life-threatening and grade 5= death related). Categories with non-zero values are presented.
Time Frame: as for outcome 2
Population: Safety analysis set included all participants who received at least one dose of study drug (avelumab or axitinib). Participants were classified according to the study treatment received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number; unit: Percentage of participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 18
Percentage of participants
  Alanine aminotransferase increased (Grade 3) | 7.3 | 5.6
  Alkaline phosphatase increased (Grade 3) | 2.4 | 11.1
  Aspartate aminotransferase increased (Grade 3) | 2.4 | 5.6
  Blood bilirubin increased (Grade 3) | 2.4 | 0
  Creatinine increased (Grade 3) | 2.4 | 5.6
  GGT increased (Grade 3): number analyzed (Participants) | 40 | 16
  GGT increased (Grade 3) | 7.5 | 18.8
  Hyperglycemia (Grade 3) | 4.9 | 5.6
  Hyperglycemia (Grade 4) | 2.4 | 0
  Hyperkalemia (Grade 3) | 7.3 | 0
  Hypermagnesemia (Grade 3) | 2.4 | 0
  Hypermagnesemia (Grade 4) | 0 | 5.6
  Hypoalbuminemia (Grade 3) | 0 | 5.6
  Hypocalcemia (Grade 3) | 4.9 | 5.6
  Hypoglycemia (Grade 4) | 2.4 | 0
  Hypokalemia (Grade 3) | 4.9 | 0
  Hypomagnesemia (Grade 3) | 2.4 | 0
  Hypomagnesemia (Grade 4) | 2.4 | 0
  Hyponatremia (Grade 3) | 9.8 | 16.7
  Hyponatremia (Grade 4) | 2.4 | 0
  Hypophosphatemia (Grade 3) | 4.9 | 5.6
  Lipase increased (Grade 3): number analyzed (Participants) | 39 | 16
  Lipase increased (Grade 3) | 10.3 | 6.3
  Lipase increased (Grade 4): number analyzed (Participants) | 39 | 16
  Lipase increased (Grade 4) | 2.6 | 6.3
  Serum amylase increase (Grade 3): number analyzed (Participants) | 40 | 16
  Serum amylase increase (Grade 3) | 2.5 | 12.5

5. Secondary Outcome: Time to Tumor Response (TTR) in Participants With Confirmed CR or PR
Description: TTR was defined as the time from the first dose of study treatment to the first documentation of objective tumor response documented in participants with confirmed objective response (CR or PR). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of start of treatment until date of first documentation of objective tumor response (maximum up to 56 months)
Population: Full Analysis Set included all participants who received at least one dose of avelumab and axitinib. Participants were classified according to the study treatment received. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 13 | 2
Months | 1.9 [1.8 to 5.3] | 2.8 [1.8 to 3.7]

6. Secondary Outcome: Duration of Response in Participants With Confirmed CR or PR
Description: Duration of response was defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first in participants with confirmed objective response (CR or PR). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first (maximum up to 56 months)
Population: Full Analysis Set included all participants who receive at least one dose of avelumab and axitinib. Participants were classified according to the study treatment received. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 13 | 2
Months | 7.5 [3.7 to 15.5] | 17.4 [5.6 to 29.2]

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from first dose of study treatment (ie, start date) to the date of progression of disease (PD) by RECIST v 1.1 or death due to any cause, whichever occurred first. PFS data was censored on the date of the last adequate tumor assessment for participants without an event (PD or death), for participants who started new anti-cancer treatment prior to an event, or for participants with an event after two or more missing tumor assessments. PD as per RECIST v1.1 for target lesions was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm. For non-target lesions PD was defined as unequivocal progression of pre-existing lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From start of study treatment until first documentation of PD or death due to any cause or censoring date (maximum of 24 months)
Population: Full Analysis Set included all participants who receive at least one dose of avelumab and axitinib. Participants were classified according to the study treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 20
Months | 5.5 [2.5 to 7.0] | 2.3 [1.8 to 5.6]

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of first study treatment to the date of death due to any cause. Participants last known to be alive were censored at date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of start of study treatment until date of death or censoring date (maximum up to 56 months)
Population: Full Analysis Set included all participants who received at least one dose of avelumab and axitinib. Participants were classified according to the study treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 20
Months | 15.4 [8.0 to 26.9] | 16.8 [2.3 to 35.4]

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Avelumab
Time Frame: Pre-dose, 1 hour post-dose on Cycle 1 Day 1, Day 15 and Cycle 2 Day 1
Population: The Pharmacokinetic (PK) parameter analysis set is a subset of the safety analysis set and included all participants who have at least one of the PK parameters of interest for avelumab or axitinib. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 35 | 15
Microgram per milliliter
  Cycle 1 (Day 1): number analyzed (Participants) | 35 | 12
  Cycle 1 (Day 1) | 235.0 (26) | 206.3 (27)
  Cycle 1 (Day 15): number analyzed (Participants) | 32 | 15
  Cycle 1 (Day 15) | 264.0 (34) | 163.9 (211)
  Cycle 2 (Day 1): number analyzed (Participants) | 29 | 15
  Cycle 2 (Day 1) | 283.2 (24) | 260.4 (25)

10. Secondary Outcome: Cmax of Axitinib
Time Frame: Pre-dose, 2 hour post-dose on Cycle 1 Day 15, Cycle 2 Day 1 and 15
Population: PK parameter analysis set is a subset of the safety analysis set and included all participants who have at least one of the PK parameters of interest for avelumab or axitinib. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 16 | 5
Microgram per milliliter
  Cycle 1 (Day 15): number analyzed (Participants) | 12 | 5
  Cycle 1 (Day 15) | 17.29 (198) | 14.64 (448)
  Cycle 2 (Day 1): number analyzed (Participants) | 16 | 3
  Cycle 2 (Day 1) | 16.46 (91) | 5.206 (448)
  Cycle 2 (Day15): number analyzed (Participants) | 10 | 4
  Cycle 2 (Day15) | 10.64 (223) | 2.868 (24)

11. Secondary Outcome: Pre-dose Observed Serum Concentration (Ctrough) of Avelumab
Time Frame: Pre-dose on Cycle 1 Day 1, 15, Cycle 2 Day 1, Cycle 3 Day 15, Cycle 6 Day 15, Cycle 9 Day 15, and Cycle 12 Day 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 39 | 19
Microgram per milliliter
  Cycle 1 (Day 1): number analyzed (Participants) | 38 | 19
  Cycle 1 (Day 1) | 0 (0) | 0 (0)
  Cycle 1 (Day 15): number analyzed (Participants) | 39 | 18
  Cycle 1 (Day 15) | 19.46 (80) | 18.84 (101)
  Cycle 2 (Day 1): number analyzed (Participants) | 32 | 17
  Cycle 2 (Day 1) | 20.96 (119) | 19.62 (91)
  Cycle 3 (Day 15): number analyzed (Participants) | 21 | 9
  Cycle 3 (Day 15) | 28.22 (55) | 39.29 (36)
  Cycle 6 (Day 15): number analyzed (Participants) | 17 | 6
  Cycle 6 (Day 15) | 29.68 (52) | 43.30 (57)
  Cycle 9 (Day 15): number analyzed (Participants) | 12 | 3
  Cycle 9 (Day 15) | 32.84 (29) | 42.41 (47)
  Cycle 12 (Day 15): number analyzed (Participants) | 6 | 3
  Cycle 12 (Day 15) | 36.71 (50) | 39.01 (20)

12. Secondary Outcome: Ctrough of Axitinib
Time Frame: Pre-dose on Cycle 1 Day 15, Cycle 2 Day 1 and 15
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 29 | 14
Microgram per milliliter
  Cycle 1 (Day 15): number analyzed (Participants) | 29 | 12
  Cycle 1 (Day 15) | 7.923 (127) | 4.613 (231)
  Cycle 2 (Day 1): number analyzed (Participants) | 28 | 14
  Cycle 2 (Day 1) | 8.871 (123) | 5.247 (172)
  Cycle 2 (Day 15): number analyzed (Participants) | 23 | 12
  Cycle 2 (Day 15) | 6.455 (129) | 3.944 (172)

13. Secondary Outcome: Number of Participants With Programmed Death-Ligand 1 (PD-L1) Status
Description: PD-L1 status was defined as positive when PD-L1 staining of any intensity was observed in >= 1% of the tumor cells. PD-L1 status was defined as negative when PD-L1 staining of any intensity was observed in < 1% of the tumor cells.
Time Frame: Screening, up to 28 days prior to Day 1
Population: Biomarker analysis set is a subset of the safety analysis set and included participants who had at least one baseline biomarker assessment. Analysis sets was defined separately for blood-based and tumor tissue-based biomarkers. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 32 | 16
Participants
  PD-L1 positive | 8 | 5
  PD-L1 negative | 24 | 11

14. Secondary Outcome: Tumour Mutational Burden (TMB) in Tumor Tissue
Description: Mutational load within tumor tissue was defined as number per megabase of the genome, coding, base substitution, and indel mutations present in the sample. Mutational load was determined in whole blood samples using next generation deoxyribonucleic acid (DNA) sequencing followed by computational analysis.
Time Frame: Screening, up to 28 days prior to Day 1
Population: Biomarker analysis set is a subset of the safety analysis set and included participants who had at least one baseline biomarker assessment. Analysis sets was defined separately for blood-based and tumor tissue-based biomarkers. Here, 'Number Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Mutations per megabase
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 24 | 15
Mutations per megabase | 2.8 (2.97) | 3.7 (4.53)

15. Secondary Outcome: T-cell Receptor (TCR) Sequencing to Identify Fraction Productive of Cells
Description: The immune response was measured by total T cell receptor (TCR) sequencing in peripheral blood and determined the characterization of immune repertoires. Fraction productive of cells is defined as the number of T cells within the total nucleated cell count (T cells and non-T cells).
Time Frame: Screening, up to 28 days prior to Day 1
Population: Biomarker analysis set is a subset of the safety analysis set and included participants who have at least one baseline biomarker assessment. Analysis sets was defined separately for blood-based and tumor tissue-based biomarkers. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Proportion of T cells
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 15 | 10
Proportion of T cells | 0.2 (0.17) | 0.1 (0.08)

16. Secondary Outcome: T-cell Receptor (TCR) Sequencing to Identify Simpson Clonality
Description: The immune response was measured by TCR sequencing in peripheral blood and determined the characterization of immune repertoires. Simpson clonality is calculated for a sample as the square root of Simpson's diversity index for all productive rearrangements. Values for clonality ranged from 0 to 1. Values near 1 represented samples with one or a few predominant rearrangements (monoclonal or oligoclonal samples) dominating the observed repertoire. Clonality values near 0 represented more polyclonal samples.
Time Frame: Pre-dose on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 15 | 10
Index | 0.1 (0.04) | 0.1 (0.03)

17. Secondary Outcome: T-cell Receptor (TCR) Sequencing to Identify Total T Cells
Description: The immune response was measured by total TCR sequencing in peripheral blood and determined the characterization of immune repertoires.
Time Frame: Pre-dose on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Cells
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 15 | 10
Cells | 1623.7 (1971.39) | 1168.4 (1450.51)

18. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) and Neutralizing Antibodies (nAb) Against Avelumab
Description: ADA and nAb positive was defined as presence of at least one positive ADA and nAb sample, respectively. NAb analysis was planned to be conducted for ADA positive samples.
Time Frame: Within 2 hours pre-dose on Cycle 1 Day 1,15, Cycle 2 Day 1; Day 15 of Cycle 3, 6, 9, 12, end of treatment and 30 days after last dose of study treatment (maximum up to 56 months)
Population: Immunogenicity analysis set is a subset of the safety analysis set and included participants who had at least one ADA assessment collected for avelumab. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows. Due to the low observed rate of the treatment-induced immunogenicity responses, none of the ADA positive samples was tested for the NAb assay.
Measure: Count of Participants; unit: Participants
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
Number analyzed (Participants) | 41 | 20
Participants
  ADA ever-Positive | 7 | 0
  nAb ever-Positive: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment or start of new anti-cancer treatment -1 day (maximum up to 56 months)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorised as serious in 1 subject and non-serious in another, or a subject may have experienced both SAE and non-SAE.
Arm/Group | NSCLC Avelumab + Axitinib | UC Avelumab + Axitinib
All-Cause Mortality (participants affected / at risk) | 27/41 | 11/20
Serious Adverse Events (participants affected / at risk) | 21/41 | 11/20
Other Adverse Events (participants affected / at risk) | 41/41 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Avelumab + Axitinib (N=41) | UC Avelumab + Axitinib (N=20)
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 2 | 0
Disease progression (General disorders) | 4 | 3
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Intracranial haematoma (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Avelumab + Axitinib (N=41) | UC Avelumab + Axitinib (N=20)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Adrenal insufficiency (Endocrine disorders) | 5 | 1
Hypothyroidism (Endocrine disorders) | 13 | 1
Asthenia (General disorders) | 7 | 5
Chills (General disorders) | 7 | 1
Fatigue (General disorders) | 9 | 5
General physical health deterioration (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 4 | 2
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 8 | 4
Stomatitis (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Urinary tract infection (Infections and infestations) | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 0
Alanine aminotransferase increased (Investigations) | 9 | 3
Amylase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 2
Blood corticotrophin increased (Investigations) | 4 | 0
Blood creatinine increased (Investigations) | 2 | 2
Blood thyroid stimulating hormone increased (Investigations) | 3 | 1
Blood triglycerides increased (Investigations) | 4 | 0
C-reactive protein increased (Investigations) | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Lipase increased (Investigations) | 3 | 2
Weight decreased (Investigations) | 9 | 6
Decreased appetite (Metabolism and nutrition disorders) | 14 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 7 | 1
Hypertension (Vascular disorders) | 17 | 4
Hypertensive crisis (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT03472560/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT03472560/SAP_001.pdf